CLINICAL TRIAL: NCT03044691
Title: The OneFlorida Cancer Control Alliance: Implementing the 6As in Pediatric Primary Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: confounding factors impacted the ability to fully complete the aims of this study
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB201600151; 4KB16 (Other Grant/Funding Number: Florida Department of Health); OCR15156 (Other: Universiy of Florida)
Record Dates: First submitted 2017-02-01; First posted 2017-02-07 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Clinic (No Intervention): The control group will have to complete the Adaptive Reserve and Change Process Capability Questionnaire and Clinician Survey at baseline and 9 months. Clinicians will provide their usual care related to tobacco and nicotine product use screening and cessation recommendations. Medical record of patients will be reviewed at baseline and at 6 months.
- Intervention Clinic (Experimental): Participants will be asked to complete the Youth Tobacco and Nicotine Product Questionnaire and Parent Brief Questionnaire (PBQ) using the ResearchACTS software at the point of care. A follow-up survey Youth Tobacco and Nicotine Product Primary Care survey will be administered to participants at least 30 days after their clinic visit.
  Interventions: Behavioral: ResearchACTS software

INTERVENTIONS:
Behavioral: ResearchACTS software — screen patients for tobacco and nicotine product use (using the anticipate and ask components of the 6As) by having youth complete a tobacco and nicotine use screening tool using the ResearchACTS software.
  Arms: Intervention Clinic

SUMMARY:
The primary purpose of our study is to conduct a pilot, practice-based intervention focused on increasing adherence to the 6As for youth ages 11 through 17 years. The 6As are: (1) "Anticipate" (future use), (2) "Ask" (about tobacco use), (3) "Advise" (advise the patient to quit using tobacco), (4) "Assess" (the patient's readiness to quit using tobacco), (5) "Assist" (by setting a quit date, providing materials on quitting tobacco, providing tobacco cessation medications, and referring the patient for additional services and/or counseling) , and (6) "Arrange" (by re-contacting the patient after their quit date and arranging a follow-up visit).

DETAILED DESCRIPTION:
Investigators will incorporate American Academy of Pediatrics (AAP) best practice recommendations to screen and counsel parents. The specific aims of this study are to: (1) Develop and deploy an electronic short screening tool for tobacco and nicotine product use into pediatric primary care workflow in conjunction with clinician and office staff training on the 6As and parent screening through the use of trained Clinical Practice Facilitators, clinician-engaged adaptations of the intervention to fit their practice workflow, and support for Maintenance of Certification (MOC) to engage pediatricians in implementing the best practices; (2) Gather pilot data about the effectiveness of the intervention on clinician adherence to best practices and changes in practice capacity for change, adaptive reserve, and clinician self-efficacy; and (3) Examine the congruence between documentation of the intervention in the electronic health record (EHR) and youth report of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 11-17 years old

Exclusion Criteria:

* 18 years and older

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2017-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shenkman, PhD, Principal Investigator — University of Florida; Ramzi Salloum, PhD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - University of Florida Clinics, Gainesville, Florida
  - UF Health Family Medicine and Pediatrics-Blanding, Jacksonville, Florida
  - UF Health Family Medicine and Pediatrics-Baymeadows, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Clinic | Intervention Clinic
Started | 0 | 84
Completed | 0 | 84
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data systems did not allow for the data needed for the aims of the control clinics
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Clinic | Intervention Clinic | Total
Number analyzed (Participants) | 0 | 84 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 84 | 84
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 32 | 32
  Male |  | 52 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States |  | 84 | 84

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of ResearchACTS Software in Clinical Assessment of Tobacco Use Measures
Description: During the recruitment period, investigators will observe feedback from patients and clinic staff on how the feasibility of using the ResearchACTS software to capture tobacco use measures in a clinical setting. Feasibility of the software tool will be demonstrated by the ability of patients to complete the assessment within the timeframe afforded during a clinical visit.
Time Frame: Baseline
Population: No-one was recruited into the control clinic arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Clinic | Intervention Clinic
Number analyzed (Participants) | 0 | 84
Participants
  Able to complete | 0 | 84
  Unable to complete | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Data systems did not allow for the data needed for the aims of the control clinics; therefore, zero participants were at risk.
Arm/Group | Control Clinic | Intervention Clinic
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/75
Other Adverse Events (participants affected / at risk) | 0/0 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT03044691/Prot_SAP_000.pdf